CLINICAL TRIAL: NCT00986310
Title: Efficacy of Fluoxetine in Reducing Ictal Hypoventilation in Patients With Partial Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 244486
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Uncontrolled Partial Epilepsy; Ictal Hypoventilation
Keywords: fluoxetine; epilepsy; Prozac
MeSH Terms: conditions — Epilepsy | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluoxetine (Active Comparator): Patients will be randomized to receive either 20 mg/day of fluoxetine (one pill) or placebo (one pill), to be started one week prior to the scheduled hospital admission date. The dose will be increased to two pills per day on day 1 of hospitalization bringing the total dose of fluoxetine to 40 mg/day in patients randomized to receive this medication. On the day of discharge from the hospital, the study medication will be reduced to 1 pill per day and the patient will be instructed to stop the medication one week following discharge.
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Patients will be randomized to receive either 20 mg/day of fluoxetine (one pill) or placebo (one pill), to be started one week prior to the scheduled hospital admission date. The dose will be increased to two pills per day on day 1 of hospitalization. On the day of discharge from the hospital, the study medication will be reduced to 1 pill per day and the patient will be instructed to stop the medication one week following discharge.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Subjects randomized to fluoxetine will receive 20mg/day (one pill) for one week. The dose will be increased to 40mg/day (two pills) for the duration of hospitalization for VET. The dose will be decreased to 20 mg/day (one pill) from the day of hospital discharge for one week, at which time the medication will be discontinued.
  Other Names: Prozac
  Arms: fluoxetine
Drug: Placebo — Subjects randomized to fluoxetine will receive 20mg/day (one pill) for one week. The dose will be increased to 40mg/day (two pills) for the duration of hospitalization for VET. The dose will be decreased to 20 mg/day (one pill) from the day of hospital discharge for one week, at which time the medication will be discontinued.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of fluoxetine on breathing mechanisms during seizures. Patients with partial epilepsy commonly have changes in their breathing mechanisms during seizures. These changes may increase the risk of serious side effects from seizures, including sudden unexplained death in epilepsy (SUDEP), which affects 2-10 per 1000 patients with epilepsy each year. Fluoxetine (Prozac) may help to stimulate breathing through its actions in the brain and has been shown to improve breathing changes seen with seizures in certain animals. Fluoxetine is in a class of medications called selective serotonin reuptake inhibitors (SSRIs). It works by increasing the amount of serotonin, a natural substance in the brain, at synapses, the junctions at which nerve cells in the brain communicate. Fluoxetine is currently approved by the United States Food and Drug Administration (FDA) for the treatment of patients with Major Depressive Disorder, Obsessive Compulsive Disorder, Bulimia Nervosa, Panic Disorder and Premenstrual Dysphoric Disorder.

DETAILED DESCRIPTION:
Patients who consent to participate in the study will come to the clinic one week prior to the scheduled date of hospitalization in the Epilepsy Monitoring Unit (EMU). At this visit a complete physical examination including vital signs and complete neurological examination, mental status, cranial nerves, motor examination, deep tendon reflexes, sensory examination, coordinator and gait will be performed. Baseline laboratory studies including complete blood count, serum electrolytes, renal and liver function studies and serum pregnancy test for female patients will also be performed. Study medication will be dispensed at this visit.

Patients will be randomized to receive either 20 mg/day of fluoxetine (one pill) or placebo (one pill), to be started one week prior to the scheduled hospital admission date. The dose will be increased to two pills per day on day 1 of hospitalization bringing the total dose of fluoxetine to 40 mg/day in patients randomized to receive this medication. On the day of discharge from the hospital, the study medication will be reduced to 1 pill per day and the patient will be instructed to stop the medication one week following discharge. A follow-up clinic visit for the patient will be scheduled 1 month following hospital discharge, as is the usual protocol for patients undergoing VET at our institution.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with temporal lobe epilepsy, aged 18-65.
2. Medical intractability of seizures such that VET to determine candidacy for epilepsy surgery is determined to be clinically appropriate for the patient by the primary treating epileptologist.
3. Intelligence Quotient >70.
4. Native English speaker or adequate fluency in English to provide informed consent.
5. Female patients of child-bearing potential must be using an acceptable method of contraception, including abstinence.

Exclusion Criteria:

1. Progressive neurological disease.
2. Severe depression, bipolar disease or psychosis.
3. History of suicidal ideation or intent.
4. Clinically significant concurrent medical illness, including hepatic or renal insufficiency and diabetes.
5. Pregnant or lactating women.
6. Current heavy alcohol or illicit drug use.
7. Patients already taking fluoxetine or other selective serotonin reuptake inhibitors (SSRIs).
8. Concurrent use of monoaminoxidase inhibitors, antipsychotic agents, antidepressant agents other than SSRIs or frequent use of triptan agents.
9. History of a previous allergic reaction or adverse effects with SSRIs.
10. History of serotonin syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Bateman, MD, FRCPC, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was completed and the PI has left the institution without entering the results information. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Period: Overall Study
Arm/Group | Fluoxetine | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was completed and the PI has left the institution without entering the results information. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years] — Population: The study was completed and the PI has left the institution without entering the results information. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Sex: Female, Male — Population: The study was completed and the PI has left the institution without entering the results information. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.

OUTCOME MEASURES:

1. Primary Outcome: The Primary End Point for This Study is a 50% Fluoxetine-related Reduction in the Number of Seizures With Associated Oxygen Desaturations Below 90% Compared With Placebo.
Time Frame: 6 weeks
Population: as for baseline characteristics
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Secondary End Point is, in the Group of Seizures With Desaturations Below 90%, a 30% Fluoxetine-related Improvement in the Oxygen Desaturation Nadir Relative to Placebo.
Time Frame: 6 weeks
Population: as for baseline characteristics
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was completed and the PI has left the institution without entering the results information. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Description: The study was completed and the PI has left the institution without entering the results information. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | Fluoxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
PI has left institution. Despite many attempts to contact, no response was received and results were not able to obtained nor entered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No